CLINICAL TRIAL: NCT06960603
Title: Effect of Pulp Inflammatory Mediators' Level on the Outcome of Full Pulpotomy in Teeth With Symptomatic Pulpitis
Brief Title: Pulp Inflammatory Markers and Outcome of Pulpotomy
Acronym: pulpitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Principal Investigator, Nessrin Taha, Professor, Jordan University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 462/2024; 462/2024 (Other Grant/Funding Number: Jordan university of Science and Technology)
Record Dates: First submitted 2025-04-26; First posted 2025-05-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pulpitis in Permanent Teeth; Dental Caries Extending to Pulp
Keywords: Permanent teeth; Deep caries; Reversible pulpitis; Irrevrsible pulpitis; Pulpotomy; Inflammatory mediators

STUDY DESIGN:
Intervention Model Description: Permanent teeth with deep caries reaching the dental pulp and requires full pulpotomy treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full pulpotomy using calcium silicate based material for teeth with carious pulp exposure (Experimental): The tooth with carious pulp exposure will be treated with full pulpotomy, Blood samples will be collected from the tooth for investigation of inflammatory mediator level. Calcium silicate based material will be placed over the pulp and the tooth will restored with resin composite.
  Patients symptoms will be monitored at 1 week postoperatively, the patient will score their pain levels on a scale from 0-10.
  The patients will be recalled at 6 and 12 months post procedure. The tooth will be examined for symptoms of pain, and radiographs will be taken. based on the findings it will be scored as success or failure of the pro cedure.
  this result will be corelated with the level of measure inflammatory mediators that were taken during the procedure.
  Interventions: Other: Full pulpotomy

INTERVENTIONS:
Other: Full pulpotomy — First: Cutting the coronal pulp tissue to the level of the root canal orifices. Second: Followed by taking samples of the pulpal blood Third: Placement of calcium silicate material capping over the pulp
  Other Names: Cervical pulpotomy

SUMMARY:
This is a prospective clinical study that aims to investigate the level of inflammatory mediators in the inflamed dental pulp and its potential relationship to the outcome of full pulpotomy in mature permanent teeth with carious pulp exposure.

Pulp blood samples from the teeth will be collected during treatment, MMP9 levels will be recorded using Elisa kits. The teeth will be restored and followed up at 1 week, 6 months, 1, and 2 years. The teeth will be assesses both clinically and radiographically. The procedure will be success if the tooth is asymptomatic clinically and with normal periapical findings. The relationship between MMP9 level and success of treatment will be investigated.

DETAILED DESCRIPTION:
Dental caries is one of the most common chronic diseases of adults and children. If left untreated, the disease can have a wide range of dental, medical, social, and quality of life consequences, such as pain, infection, early tooth loss, and loss of self-confidence.

Full pulpotomy is a vital pulp therapy procedure that involves the removal of the coronal pulp to the levels of canal orifices followed by achieving hemostasis and placement of a biocompatible capping material. Full pulpotomy has been proved to be a promising alternative treatment option to the conventional root canal treatment in cariously exposed molars with either diagnosis of reversible or irreversible pulpitis.

Clinically, diagnosing the actual histopathological status of the inflamed pulp is challenging and is an empirical guess based on the results of sensibility testing and patients' symptoms. In recent years there has been an attempt to investigate the level of inflammatory mediators in the pulp, with an attempt to develop a chairside diagnosis tool that will help better in diagnosing the state of the pulp; and therefore, predict the outcome of treatment procedures.

In recent years matrix metalloproteinases (MMPs) have been increasingly studied for their role in the diagnosis of dental inflammatory processes. Several studies evaluated the correlation between inflammation of the dental pulp and the levels of MMPs (MMP-1, -2, -3,-8 and -9), in addition to other molecular markers like interluekins and prostaglandins.

However, the use of concentrations of MMPs in the pulpal blood as a marker to differentiate between reversible and irreversible pulpitis has not been thoroughly investigated yet.

The aim of the study is to investigate the inflammatory mediators' level in inflamed pulps and to assess its relation to the outcome of full pulpotomy in carious teeth with symptomatic pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* Non -contributory medical history (ASA 1)

  * Molar tooth with deep caries extending>= 2/3 of dentine or exposing the pulp on the radiograph
  * The tooth should give positive response to cold sensibility testing
  * Clinical diagnosis of either reversible or irreversible pulpitis based on the symptoms and results of cold testing.
  * The tooth is restorable, probing pocket depth and mobility are within normal limits

Exclusion Criteria:

* Non-restorable tooth.

  * Signs of pulpal necrosis including sinus tract or swelling.
  * No enough bleeding after the pulpotomy procedure.
  * Inability to achieve hemostasis within 10 min after the pulpotomy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 1 week, 6 months , 12 months
  Pain levels after the procedure will be assessed on a scale from 0-10, at 1 week, 6 months an 12 months postoperatively.
  The procedure will be considered success if the tooth is symptom free and pain levels range form 0-3.
  It will be considered as a failure If pain levels are >0-3

SECONDARY OUTCOMES:
Radiographic Findings | 6, 12, 24 months
  A periapical x-ray will be taken for the tooth immediately after treatment and at 6 12, and 24 months follow up.
  For success the tooth should be free of root resorption and free of bone resorption around the root

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin A Taha, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan university of science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available upon reasonable request after officila publication and termination of recruitment

REFERENCES:
- [Background] Sharma R, Kumar V, Logani A, Chawla A, Mir RA, Sharma S, Kalaivani M. Association between concentration of active MMP-9 in pulpal blood and pulpotomy outcome in permanent mature teeth with irreversible pulpitis - a preliminary study. Int Endod J. 2021 Apr;54(4):479-489. doi: 10.1111/iej.13437. Epub 2020 Dec 13. PMID 33128238
- [Background] Taha NA, About I, Sedgley CM et al. Conservative management of mature permanent teeth with carious pulp exposure. J Endod 2020; 46: S33-S4. Taha NA, Al-Khatib H. 4-Year Follow-up of Full Pulpotomy in Symptomatic Mature Permanent Teeth with Carious Pulp Exposure Using a Stainproof Calcium Silicate-based Material. J Endod 2022; 48: 87-95. Taha NA, Al-Rawash MH, IMRAN ZA. Outcome of full pulpotomy in mature permanent molars using 3 calcium silicate-based materials: A parallel, double blind, randomized controlled trial. Int Endod J 2022; 55:416-29.
- [Background] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305